CLINICAL TRIAL: NCT05067296
Title: Prevalance of Cesarean Section Niche in Patients With Abnormal Uterine Bleeding
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Mahmoud Ramadan Hafez (Other)
Responsible Party: Sponsor-Investigator, Mahmoud Ramadan Hafez, Mahmoud Ramadan Hafez Ahmed, Sohag University
Organization: Sohag University (Other)
Other Study IDs: Soh-Med-21-09-06
Record Dates: First submitted 2021-09-23; First posted 2021-10-05 (Actual); Last update posted 2021-10-05 (Actual); Status verified 2021-09

CONDITIONS: Cesarean Section Niche and Abnormal Uterine Bleeding
MeSH Terms: conditions — Metrorrhagia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cesarean section niche and patients with abnormal uterine bleeding: Observation by Tvs
  Interventions: Other: By TVS
- Abnormal uterine bleeding in patients without Cesarean section niche: Observation by Tvs
  Interventions: Other: By TVS

INTERVENTIONS:
Other: By TVS — Uses of TVS to diagnosis of Cesarean section niche in patients with abnormal uterine bleeding

SUMMARY:
Prevalance of Cesarean section niche in patients with abnormal uterine bleeding

ELIGIBILITY:
Inclusion Criteria:

Age between 20-40 years old. Non pregnant women. Previous cesarean section (one or more). Presence of abnormal uterine bleeding

Exclusion Criteria:

Virgins Pregnant women. Patients with vaginal delivery. Patients with uterine bleeding with known cause.

Ages: 20 Years to 40 Years | Sex: Female
Age Groups: Adult
Study Population: Prevalance of Cesarean section niche in patients with abnormal uterine bleeding
Sampling Method: Non-Probability Sample
Enrollment: 1 (Estimated)
Dates: Start 2021-10-01 (Estimated); Primary Completion 2022-04-01 (Estimated); Study Completion 2022-08-01 (Estimated)

PRIMARY OUTCOMES:
Cesarean section niche in patients with abnormal uterine bleeding | 6 months
  To study relationship between the niche and the abnormal uterine bleeding

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University, Sohag, Egypt